CLINICAL TRIAL: NCT03094897
Title: Phase 1 Study of 18F-Al-NOTA-MATBBN in Cancer Diagnostics
Brief Title: Clinic Study of 18F-Al-NOTA-MATBBN in Cancer Diagnostics
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wuxi4PH
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Neoplasms; Prostatic Neoplasms
Keywords: Breast Neoplasms,Prostatic Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 18F-Al-NOTA-MATBBN PET/CT (Experimental): Imaging with 18F-Al-NOTA-MATBBN PET/CT
  Interventions: Drug: 18F-Al-NOTA-MATBBN PET/CT; Device: PET/CT

INTERVENTIONS:
Drug: 18F-Al-NOTA-MATBBN PET/CT — 18F-Al-NOTA-MATBBN(PET imaging agent) given by vein before PET scans.Perform PET/CT for each enrolled volunteer or patient at 60-90min.
Device: PET/CT — Imaging with 18F-Al-NOTA-MATBBN PET/CT.

SUMMARY:
The purpose of this study is to determine whether 18F-Al-NOTA-MATBBN is safety and effective for cancer diagnosis.

DETAILED DESCRIPTION:
Observe radiation dose to healthy volunteers and patients; the correlation between integrin level and tumor/metastases uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers or patients with age more than 18 yeas;
2. The patients have been diagnosed with cancer or suspected with cancer;
3. It must fulfill the ethical requirements and subjects have signed an informed consent.

Exclusion Criteria:

1. Pregnancy or nursing mothers;
2. Having drugs or alcohol dependence;
3. Hypersensitive to the active or inactive ingredients of the study drug;
4. Having attended other drug clinical trials within three months;
5. Cardiac functional insufficiency;
6. Hepatic and renal function insufficiency;
7. Hypertensive patients with serious complications;
8. Endangering the safety of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-20 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 18F-Al-NOTA-MATBBN in malignant lesions | 1 day
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in malignant lesions will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: chunjing Yu, PhD, Principal Investigator — Department of Nuclear Medicine, Affiliated Hospital of Jiangnan University (Wuxi 4th People's Hospital)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Honer M, Mu L, Stellfeld T, Graham K, Martic M, Fischer CR, Lehmann L, Schubiger PA, Ametamey SM, Dinkelborg L, Srinivasan A, Borkowski S. 18F-labeled bombesin analog for specific and effective targeting of prostate tumors expressing gastrin-releasing peptide receptors. J Nucl Med. 2011 Feb;52(2):270-8. doi: 10.2967/jnumed.110.081620. Epub 2011 Jan 13. PMID 21233180